CLINICAL TRIAL: NCT01161979
Title: A Randomized. Single-Dose, Two-Way Crossover Relative Bioavailability Study of Zonisamide Formulations in Normal, Healthy Men and Women Following a Standard Meal
Brief Title: Bioequivalence Study of Zonisamide Capsules 100 mg of Dr.Reddy's Laboratories Limited Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Vice president-Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 40578
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2005-01

CONDITIONS: Healthy
MeSH Terms: interventions — Zonisamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zonisamide (Experimental): Zonisamide Capsules 100 mg of Dr.Reddy's laboratories Limited
  Interventions: Drug: Zonisamide
- Zonegran (Active Comparator): Zonegran Capsules 100 mg of EISAI INC
  Interventions: Drug: Zonegran

INTERVENTIONS:
Drug: Zonisamide — Zonisamide capsules 100 mg
  Other Names: Zonegran Capsules 100 mg
  Arms: Zonisamide
Drug: Zonegran — Zonegran Capsules 100 mg of EISAI INC
  Arms: Zonegran

SUMMARY:
The objective of this study was to compare the rate and extent of absorption of Dr. Reddy's Zonisamide 100 mg Capsule to that of Zonegran® 100 mg Capsule after a single, one-capsule dose in subjects fed a high standard fat meal.

DETAILED DESCRIPTION:
This was an open label, randomized, balanced, single dose, two-period, two-treatment, two-sequence crossover study, performed under fed conditions. Subjects were confined to the SFBC Clinical Research Facility from at least 10 hours prior to drug administration, until after the 24-hour post-dose blood draw, in each period. The treatment phases were separated by a washout period of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Is the individual a healthy, normal adult man or non-child bearing potential woman who volunteers to participate?
* Is s/he at least 18 years of age?
* Is his/her BMI between 19 and 30, inclusive?
* Is s/he considered reliable and capable of understanding his/her responsibility and role in the study?
* Has s/he provided written informed consent?

Exclusion Criteria:

* Does the individual have a history of allergy or hypersensitivity to zonisamide or sulfonamides?
* Does s/he have clinically significant laboratory abnormalities that would interfere with the conduct or interpretation of the study or jeopardize his/her safety? Does s/he have significant history or clinical evidence of auto-immune, cardiovascular, gastrointestinal, hematological, hematopoietic, hepatic, neurological, ongoing infection, pancreatic, or renal diseases that would interfere with the conduct or interpretation of the study or jeopardize his/her safety?
* Does s/he have serious psychological illness?
* Does s/he have significant history (within the past year) or clinical evidence of alcohol or drug abuse?
* Does s/he have a positive urine drug screen, or a positive HIV-1, or hepatitis B or C screen, or a positive pregnancy test?
* Has s/he consumed grapefruit or grapefruit juice during the 7-day period preceding study initiation?
* Is s/he unable to refrain from the use of alcohol or xanthine-containing foods or beverages during periods beginning 48 hours prior to study drug administration and ending when the last blood sample has been taken?
* Has s/he used any prescription drug during the 14-day period prior to study initiation, or any OTC drug during the 72-hour period preceding study initiation?
* Is s/he unable to refrain from the use of all concomitant medications during the study?
* Has s/he donated or lost blood, or participated in a clinical study which involved the withdrawal of a large volume of blood (480 mL or more), during the six week period preceding study initiation?
* Has s/he donated plasma during the two week period preceding study initiation?
* Has s/he received an investigational drug during the 30 day Period preceding study initiation?

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-01; Primary Completion 2005-02 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence on Cmax,AUC and Tmax Parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio R Pizarro, M.D, Principal Investigator — SFBC Ft. Myers, Inc
Locations (1):
- SFBC Ft. Myers, Inc., Fort Myers, Florida, United States